CLINICAL TRIAL: NCT01677325
Title: The Clinical Trail Of NAFLD Treated By Traditional Chinese Medicine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Wen-Jian Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-65
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: NAFLD( Non-alcoholic Fatty Liver Disease )

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chinese herb (Experimental): Chinese herb
  Interventions: Drug: Chinese herb (YiQiSanJu)

INTERVENTIONS:
Drug: Chinese herb (YiQiSanJu) — Chinese herb formula:Huangqi,huanglian,yinchen,ect
  Other Names: YiQiSanJu Formula

SUMMARY:
To investigate in subjects with non-alcoholic fatty liver disease the direct effects of a Chinese herb formula.

DETAILED DESCRIPTION:
1) Liver fat (measured by CT scan) and liver function assessed by liver enzymes levels; 2) Insulin sensitivity measured by HOMA index, oral glucose tolerance test (OGTT) and a euglycaemic hyperinsulinaemic clamp (with stable isotopes) in a subset of the subjects; 3) Plasma lipid profile and non esterified fatty acids (NEFA) concentration; 4) Circulating levels of adipokines.

ELIGIBILITY:
Inclusion Criteria:

* subjects with NAFLD(nonalcoholic fatty liver disease) (criteria of Society of Hepatology, Chinese Medical Association, 2002.10),
* aged 18-65
* alcohol consumption less than 40g/week;
* liver/spleen (L/S) ratio no more than 1 by CT scan.

Exclusion Criteria:

* ALT more than twice the upper end of the normal range
* viral hepatitis
* total parenteral alimentation or secondary liver disease such as hepatocirrhosis, autoimmune hepatitis, metabolic liver disease or drug induced liver disease
* severe cardiovascular or renal dysfunction
* Subjects with diabetes (fasting glucose more than or equal to 7.0mmol/L or postprandial glucose more than or equal to 11.1mmol/L)
* Subjects treated with statins

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The CT ratio of liver/spleen | 12 weeks
  CT imaging has been used to assess hepatic steatosis and has been validated in relation to liver biopsy .The ratio of liver to spleen (L/S ratio) for CT attenuation values is an index, with a L/S ratio<1 considered to represent fatty liver .

SECONDARY OUTCOMES:
BMI(Body Mass Index ) | 12 weeks
  Body Mass Index,(weight/height^2)
liver function | 12 weeks
  Liver function enzymes- alanine aminotransferase (ALT,U/L), aspartate aminotransferase (AST,U/L) and γ-glutamyltransferase (GGT,U/L) and total bilirubin (TBI,μmol/L), albumin/globin (A/G)(Automatic biochemical analyzer)
lipid profile | 12 weeks
  Plasma lipids including triglyceride (TG,mmol/L), total cholesterol, low-density lipoprotein (LDL.mmol/L), high-density lipoprotein (HDL,mmol/L), apolipoprotein A (ApoA,mmol/L), apolipoprotein B (ApoB,mmol/L) and lipoprotein (a) (Lp(a),mmol/L). (Automatic biochemical analyzer)
NEFA(nonesterified fatty acid) | 12 weeks
  Insulin sensitivity of lipolysis using NEFA concentrations(μmol/L).(Enzyme-linked immunosorbent assay)
HOMA index | 12 weeks
  HOMA index(FBG*INSULIN/22.5)
adiponectin | 12 weeks
  adiponectin(pg/ml,Enzyme-linked immunosorbent assay)
IL-6(interleukin 6) | 12 weeks
  interleukin 6(pg/ml,Enzyme-linked immunosorbent assay)
hs-CRP (C-reactive protein) | 12 weeks
  high sensitivity C-reactive protein(mg/L,Enzyme-linked immunosorbent assay)
TNFα( tumor necrosis factor-α) | 12 weeks
  tumor necrosis factor-α(ng/L,Enzyme-linked immunosorbent assay)
leptin | 12 weeks
  leptin(ng/ml,Enzyme-linked immunosorbent assay)

OTHER OUTCOMES:
renal function | 12 weeks
  creatinine(umol/L) ,usea nitrogen(mmol/l) and uric acid(umol/L)(Automatic biochemical analyzer)
Routine blood | 12 weeks
  automatic blood analyzer. White Blood Cell Count:/L; Red Blood Cell Count:/L; Hemoglobin:g/L; Platelets:/L; neutrophilic granulocyte:％.
Routine urine examination | 12 weeks
  automatic urine analyzer. Color,odor,specific gravity,pH,Protein(g/L),Glucose(+-).
Routine stool examination | 12 weeks
  automatic stool analyzer. Color, white blood cell(/Visual Fields), red blood cell(/Visual Fields), bacteria(/Visual Fields),occult blood(+-)
electrocardiography | 12 weeks
  automatic electrocardiograph machine
chest x-ray check | 12 weeks
  diagnostic X-ray apparatus

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jian Wang, Ph.D,MD, Principal Investigator — Huashan Hospital, affliated to Fudan University